CLINICAL TRIAL: NCT05816525
Title: The Prognostic Impact of Symptoms and Lesion Depth in Partial Removal of Carious Tissue
Status: Recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Katri Croft, Principal Investigator, DDS, Specialist in Clinical Dentistry (Cariology and Endodontology), PhD candidate, University of Helsinki
Other Study IDs: PARTIALCARIESREMOVAL
Record Dates: First submitted 2023-03-27; First posted 2023-04-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Deep Caries; Pulpitis Reversible; Pulp Hyperemia
Keywords: vital pulp therapy; deep carious lesion; selective carious tissue removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Partial removal of carious tissue — Nonselective carious tissue excavation will be performed in the periphery of the cavity to achieve a good marginal seal. In the pulpal wall selective, partial carious tissue excavation is performed to the soft dentin, removing tissue only the amount that is necessary for placing the restoration. The tooth is restored with high-viscosity glass-ionomer cement.
Procedure: Final restoration — The teeth will be restored with composite resin after 12 months follow up, if the tooth is asymptomatic, responds to sensibility tests and there are no periapical changes radiographically. Glass ionomer cement will be only partially removed to create space for the final restoration.

SUMMARY:
The goal of this prospective, observational clinical cohort study is to study the effect of the preoperative condition of the tooth on the outcome of partial removal of carious tissue in mature teeth in adults. The main questions the study aims to answer are:

* Do preoperative symptoms affect the outcome?
* Does the depth of the carious lesion affect the outcome?

One hundred participants will be recruited. Patients who meet the eligibility criteria will be asked to give their informed consent to participate in the study. Partial carious tissue removal will be performed regardless of participation in the study because selective carious tissue removal is the standard treatment of choice for a vital tooth with a deep carious lesion according to the Finnish national treatment guidelines. Participants will be asked to fill in a questionnaire regarding symptoms 7 days post-treatment. The teeth will then be followed up for 12-24 months.

The null hypothesis is that there is no difference in the success between i) deep and extremely deep carious lesions and ii) initial and mild pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* the patient is communicating in the Finnish or English language
* a deep primary or secondary carious lesion in 1st or 2nd premolar or molar on occlusal or proximal surface, extending to the deepest quarter of dentine assessed from the radiograph
* asymptomatic or symptoms not more severe than reversible pulpitis (mild pulpitis according to the new pulpitis classification proposal)
* pulp responding to the electric pulp testing and cold testing
* the periodontal stage of the tooth should be I or II.

In case the patient has several teeth fulfilling the inclusion criteria, the one with the deepest lesion and/or most severe symptoms is chosen to the study.

Exclusion Criteria:

* general medical condition which makes the patient more susceptible to odontogenic infection complications
* pregnancy, breastfeeding
* mental retardation, memory disorder
* the carious lesion is extending to more than three surfaces or to both proximal surfaces
* the tooth has previous other filling(s): i) extending deeper than to the outer third of dentine; or ii) the filling is larger than Class I or II; or iii) Class II filling is not restricted to enamel; or iv) the filling has secondary/residual caries
* the tooth is not restorable
* periapical changes in the periapical radiograph
* sensitivity to percussion; swelling; sinus tract; increased mobility; resorption
* furcal lesion more severe than Class I
* ongoing orthodontic treatment
* declining to sign the written consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The first 100 consecutive patients that have entered the dental clinics involved, fulfilling the inclusion criteria, have given their informed consent, and have responded to the questionnaire after 7 days post-treatment, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success at the follow up | 12-24 months
  Symptoms and the clinical condition of the tooth will be evaluated at the follow up. In particular, the response of the tooth to both cold and EPT will be tested. In addition, a periapical radiograph will be taken. An asymptomatic tooth that responds positively to sensibility testing (both cold and EPT) and has no signs of infection clinically or in a periapical radiograph, is considered a success.

SECONDARY OUTCOMES:
Symptoms 7 days post-treatment | 7 days
  The participants will be asked to fill in an electronic questionnaire 7 days after the partial carious tissue removal. The participants will be asked whether the tooth was asymptomatic or symptomatic i) pre-treatment and ii) on the day of treatment after local anesthesia, iii) 3 days post-treatment and iv) 7 days post-treatment. Multi-choice questions will be used to find out about the nature and intensity of pain.
Pain severity using Visual Analogue Scale (VAS) 7 days post-treatment | 7 days
  The participants will be asked to fill in an electronic Visual Analogue Scale (VAS) 7 days after the partial carious tissue removal. VAS will be used to assess the severity of pain experienced. The scale will be 0-10, 0 indicating no pain and 10 indicating worst pain imaginable. The participants will be asked about pain severity i) pre-treatment, ii) on the day of treatment after local anesthesia, iii) 3 days post-treatment and iv) 7 days post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Uusimaa Wellbeing Services County, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolters WJ, Duncan HF, Tomson PL, Karim IE, McKenna G, Dorri M, Stangvaltaite L, van der Sluis LWM. Minimally invasive endodontics: a new diagnostic system for assessing pulpitis and subsequent treatment needs. Int Endod J. 2017 Sep;50(9):825-829. doi: 10.1111/iej.12793. No abstract available. PMID 28776717